CLINICAL TRIAL: NCT01493011
Title: A Randomized Contrasted Polycentric Clinical Study About Chemotherapy Combined With Whole-body Hyperthermia(WBH)to Treat Stage IIIB/IV Non Small Cell Lung Cancer (NSCLC)
Brief Title: Chemotherapy Combined With Whole-body Hyperthermia to Treat Stage IIIB/IV Non Small Cell Lung Cancer
Acronym: WBH&NSCLC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FMMU
Record Dates: First submitted 2011-12-07; First posted 2011-12-15 (Estimated); Last update posted 2012-05-15 (Estimated); Status verified 2012-05

CONDITIONS: Non-small Cell Lung Cancer Stage IIIB; Toxicity Due to Chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Drug Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- chemotherapy & WBH (Experimental): Standard chemotherapy protocol combined with whole body hyperthermia
  Interventions: Device: chemotherapy & WBH
- chemotherapy (No Intervention): standard chemotherapy protocol for advanced NSCLC

INTERVENTIONS:
Device: chemotherapy & WBH — standard first-line chemotherapy combined with whole-body hyperthemia to treat stage Ⅲb/Ⅳ NSCLC
  Arms: chemotherapy & WBH

SUMMARY:
Millions of patients die of non-small cell lung cancer (NSCLC) every year. There are several methods to treat NSCLC, including surgery, chemotherapy, radiotherapy and bioimmuotherapy. Recently, hyperthermia therapy has played an important role in neoplasm therapy. It has showed some effect in NSCLC both in animal experiment and clinical practice, yet there is little literature about Whole-body Hyperthermia (WBH) with neoplasm. The investigators decides to develop this randomized contrasted multicenter clinical study to testify to the effect of chemotherapy combined with WBH to treat stage IIIB/IV Non Small Cell Lung Cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

1. Older than 18, survive more than 3 months;
2. Pathologically or cytologically proven stage IIIB/IV non small cell lung cancer(NSCLC);
3. Measurable disease, defined as lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 2 cm with conventional techniques or as ≥ 1 cm with spiral CT scan No known CNS tumors, including brain metastases;
4. ECOG performance status 0-2;
5. Granulocytes ≥ 1,500/μL Platelets ≥ 75,000/μL Hemoglobin ≥ 8.5 g/dL Bilirubin ≤ 3 mg/dL ALT and AST ≤ 2 times upper limit of normal (ULN) PT/INR ≤ 1.7 (therapeutic anticoagulation [e.g., coumadin or heparin] allowed provided there is no prior evidence of underlying abnormality in these parameters) Creatinine ≤ 1.5 times ULN OR creatinine clearance ≥ 60 mL/min;
6. Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception before, during, and for 30 days after completion of study therapy;
7. Other prior adjuvant therapy is allowed provided it was completed > 6 months ago AND there is documented recurrence of NSCLC;
8. No prior local therapy for the target lesion unless the target lesion located within the field of local therapy has shown ≥ 25% increase in size since last treatment;
9. At least 4 weeks since prior and no concurrent palliative radiotherapy No concurrent combination anti-retroviral therapy for HIV;
10. volunteers who signed informed consent.

Exclusion Criteria:

1. During Screening period and treatment period, the main target for lesions has been given radiation;
2. The body has metal material, including a metal JieYuHuan/support/operation fixed material within;
3. Existing cerebrovascular diseases and central nervous system tumors, including metastatic carcinoma;
4. Patients with recent or ongoing gastrointestinal bleed may not be transfused to reach the entry hemoglobin of 8.5 g/dL Physicians should ensure patients requiring transfusion prior to registration do not have an occult or clinically apparent gastrointestinal bleed No history of bleeding diathesis;
5. No significant history of cardiac disease, including any of the following: NYHA class III-IV congestive heart failure Myocardial infarction within the past 6 months Cardiac arrhythmias requiring anti-arrhythmic therapy (other than beta blockers or digoxin) LVEF < 45% (or below the normal limit at the individual institution) by scintigraphy (MUGA or myocardial scintigram) History of hypertension allowed provided it is well controlled (i.e., BP < 140/90 mm Hg) on a regimen of anti-hypertensive therapy
6. Other prior adjuvant therapy is allowed provided it was completed > 6 months ago AND there is documented recurrence of NSCLC
7. No prior systemic therapy for metastatic disease At least 4 weeks since prior locoregional therapy (e.g., embolization, chemoembolization [except with doxorubicin hydrochloride], radiotherapy, or radioactive microspheres)
8. No prior local therapy for the target lesion unless the target lesion located within the field of local therapy has shown ≥ 25% increase in size since last treatment
9. poor Compliance, not receiving medication or follow-up according to study plan;
10. There are other serious situations contrary to the scheme
11. Existing tuberculosis;
12. Exist two or multiple tumors

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2011-11; Primary Completion 2012-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | one year

SECONDARY OUTCOMES:
Toxicity as assessed by NCI CTC v3.0 | one year
overall suivival | one year
quality of life | one year
Disease Control Rate | one year

CONTACTS AND LOCATIONS:
Overall Officials: LIU WENCHAO, PROFESSOR, Study Chair — xijing hospital of the fourth military medical univercity
Locations (1):
- Xijing Hospital, Xi’an, Shanxi, China